CLINICAL TRIAL: NCT00945217
Title: Genetic Probes of Atherogenic Dyslipidemia: The Roles of the SAH Gene Family (Study 2. Postmenopausal Women)
Brief Title: The Roles of SAH Gene Family in Athrogenic Dyslipidemia in Postmenopausal Women
Acronym: MOSAH-S2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Attending Physician, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 98-01-63A
Record Dates: First submitted 2009-04-17; First posted 2009-07-24 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Disorder Associated With Menstruation and/or Menopause; Dyslipidemia
Keywords: Atherogenic dyslipidemia; Non-HDL-C; Postmenopausal women; SAH gene family
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples With DNA - samples retained, with potential for extraction of DNA from buffy coats
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postmenopausal women: women with natural menopause

SUMMARY:
Atherogenic dyslipidemia is characterized by high levels of apolipoprotein B (apoB)-containing lipoproteins, including very-low-density lipoprotein (VLDL) and its remnants and small, dense LDL (sdLDL) particles, and reduced levels of high-density lipoprotein cholesterol (HDL-C). The National Cholesterol Education Program (NCEP) recommended using non-high-density lipoprotein cholesterol (non-HDL-C) to surrogate atherogenic lipoproteins in clinical practice. Recently, the investigators have done a pilot study to study the associations between SAH gene variants and atherogenic dyslipidemia (surrogated by non-HDL-C) in postmenopausal women. The investigators found that homozygosity for SAH haplotype 3 was associated with increased adiposity, insulin resistance, and elevated levels of non-HDL-C in the postmenopausal women. Based on the findings of the pilot study, the investigators plan to expand the cohort of postmenopausal women to about 800 women, that is, recruited 660 new subjects in two years. The associations between non-HDL-C and the SAH gene family will be done. Fasting blood sampling for buffy coats and lipids is the core test of Study 2. A 75-g oral glucose tolerance test (OGTT) will be available as an optional test for a better phenotyping of insulin resistance for the participants. Detailed lipid profiling including measurements of VLDL cholesterol, VLDL-TG, remnant lipoprotein, LDL particle size, apoA1, apoB, and apoCIII will be done in the second year of the study if significant associations between gene variants of the SAH gene family and non-HDL-C are detected.

DETAILED DESCRIPTION:
Atherogenic dyslipidemia is characterized by high levels of apolipoprotein B (apoB)-containing lipoproteins, including very-low-density lipoprotein (VLDL) and its remnants and small, dense LDL (sdLDL) particles, and reduced levels of high-density lipoprotein cholesterol (HDL-C). Extensive evidence shows that atherogenic dyslipidemia contributes not only to residual macrovascular risk but also to inflammation and microvascular complications. The National Cholesterol Education Program (NCEP) recommended using non-high-density lipoprotein cholesterol (non-HDL-C) to surrogate atherogenic lipoproteins in clinical practice. Elevated non-HDL-C may represent abnormal secretion, abnormal catabolism, and/or abnormal hepatic uptake of triglycerides (TG)-rich lipoproteins. Recently, we have done a pilot study to study the associations between SAH gene variants and atherogenic dyslipidemia (surrogated by non-HDL-C) in postmenopausal women. We found that homozygosity for SAH haplotype 3 was associated with increased adiposity, insulin resistance, and elevated levels of non-HDL-C in the postmenopausal women. Moreover, researchers have identified that there are at least four members in the SAH gene family: SAH, MACS1, MACS2, and MACS3. All of them seem to have acyl-CoA synthetase activity toward medium-chain fatty acids and all are clustered in chromosome 16p12. In the present study, we propose to do a two-year study to examine the associations between the SAH gene family and atherogenic dyslipidemia in postmenopausal women.

Based on the findings of the pilot study, we plan to expand the cohort of postmenopausal women to about 800 women, that is, recruited 660 new subjects in two years. The associations between non-HDL-C and the SAH gene family will be done 18 months after the study started. Fasting blood sampling for buffy coats and lipids is the core test of Study 2. A 75-g oral glucose tolerance test (OGTT) will be available as an optional test for a better phenotyping of insulin resistance for the participants. Detailed lipid profiling including measurements of VLDL cholesterol, VLDL-TG, remnant lipoprotein, LDL particle size, apoA1, apoB, and apoCIII will be done in the second year of the study if significant associations between gene variants of the SAH gene family and non-HDL-C are detected.

ELIGIBILITY:
Inclusion Criteria:

* Naturally postmenopausal women
* Not menstruated within the last 12 months.
* Willing to participate by signing an informed consent

Exclusion Criteria:

* Patients of known history of type 2 diabetes.
* Those with fasting glucose ≥ 126 mg/dL.
* History of major renal, liver, heart, and neurological disease.
* History of hyperthyroidism or hypothyroidism.
* History of acute illness in the past 6 months.
* History of alcoholism or drug abuse.
* Women who are pregnant.
* Current or concomitant illness that would interfere with the subject's ability to perform the study or that would confound the study results, judged by the investigation physicians.
* Any concomitant medication within 2 weeks of the study.
* Difficult venous access

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers with natural menopause from a research clinic
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2009-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
the differences in haplotype frequencies of the SAH gene between two groups of subjects with different levels of non-HDL-C. | 2 years

SECONDARY OUTCOMES:
the differences in haplotype frequencies of other members of the SAH gene family between two groups of subjects with different levels of non-HDL-C. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Section of Endocrinology and Metabolism, Department of Medicine, Taipei Veterans General Hospital, Taipei, Taiwan